CLINICAL TRIAL: NCT03604692
Title: A Phase 1/2, Open-Label, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamic Activity, and Efficacy of SNDX- 6352 in Subjects With Active Chronic Graft Versus Host Disease Who Have Received at Least 2 Lines of Prior Therapy
Brief Title: A Phase 1/2 Study to Evaluate Axatilimab in Participants With Active cGVHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-6352-0503
Record Dates: First submitted 2018-07-10; First posted 2018-07-27 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Chronic Graft-versus-host-disease
Keywords: cGVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — axatilimab

STUDY DESIGN:
Intervention Model Description: The dose-escalation phase is a sequential group (dose-escalating) treatment study that is open-label. The dose-expansion phase is a parallel group treatment study with open-label cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohorts of escalating dose levels of axatilimab (Experimental): Escalating dose levels of axatilimab to establish the optimal biologic dose (OBD) and recommended Phase 2 dose (RP2D).
  Intravenous (IV) infusion; axatilimab at a dose of 0.15 milligrams (mg)/kilogram (kg) to 3 mg/kg.
  Interventions: Drug: axatilimab
- Phase 2 Dose Expansion (Experimental): Phase 2, dose expansion, is an open-label design, evaluating the 1 mg/kg dose in a larger sample size.
  IV infusion; axatilimab at a dose of 1 mg/kg.
  Interventions: Drug: axatilimab

INTERVENTIONS:
Drug: axatilimab — axatilimab is a high affinity antibody targeting the colony stimulating factor 1 receptor (CSF-1R). CSF-1R signaling has been demonstrated in nonclinical studies to be the key regulatory pathway involved in the expansion and infiltration of donor derived macrophages that mediate the disease processes involved in cGVHD.
  Other Names: Niktimvo; SNDX-6352

SUMMARY:
This is a Phase 1/2, Open-label, Dose Escalation study to investigate axatilimab in participants with active chronic graft versus host disease (cGVHD).

DETAILED DESCRIPTION:
This is a dose escalation and dose expansion study in participants with active cGVHD who have received at least 2 lines of prior therapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant must be 6 years of age or older, at the time of signing the informed consent.
2. Participants who are allogeneic hematopoietic stem cell transplant (HSCT) recipients with cGVHD requiring systemic immune suppression.
3. Participants with active cGVHD who have received at least 2 lines of therapy. Participants 18 or older with active cGVHD who have erythematous rash involving >25% body surface area or a NIH mouth score of >4 must have received prior ibrutinib therapy.

   a. Active cGVHD is defined as the presence of signs and symptoms of cGVHD per 2014 NIH Consensus Development Project on Criteria for Clinical trials in cGVHD.
4. Participants may have persistent active acute and cGVHD manifestations (overlap syndrome), as defined by 2014 NIH Consensus Development Project on Criteria for Clinical trials in cGVHD.
5. Karnofsky Performance Scale of ≥60 with a life expectancy of at least 3 months (if aged 16 years or older); Lansky Performance Score of ≥60 (if less than 16 years).
6. Adequate organ and bone marrow functions.
7. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
8. Capable of giving signed informed consent which includes compliance with the study requirements and restrictions.

Key Exclusion Criteria:

1. Has acute GVHD without manifestations of cGVHD.
2. Any evidence (histologic, cytogenetic, molecular, hematologic, or mixed) of relapse of the underlying cancer or post-transplant lymphoproliferative disease at the time of screening.
3. History or other evidence of severe illness, uncontrolled infection or any other conditions that would make the participant, in the opinion of the Investigator, unsuitable for the study.
4. Known history of human immunodeficiency virus (HIV) or active hepatitis C virus (HCV) or hepatitis B virus (HBV).
5. Diagnosed with another malignancy (other than malignancy for which transplant was performed) within 3 years of enrollment, unless previously treated with curative intent and must be approved by Sponsor medical monitor (for example, completely resected basal cell or squamous cell carcinoma of the skin, resected in situ cervical malignancy, resected breast ductal carcinoma in situ, or low-risk prostate cancer after curative resection).
6. Female participants who are pregnant or breastfeeding.
7. Previous exposure to study intervention or known allergy/sensitivity to study intervention.
8. Taking agents other than a corticosteroid and one calcineurin inhibitor (CNI) for treatment of cGVHD (This does not include agents being prescribed expressly for the treatment of acute GVHD).
9. Receiving an investigational treatment within 28 days of study entry.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2024-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vedran Radojcic, M.D., Study Director — Syndax Pharmaceuticals
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Utah Health Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kitko CL, Arora M, DeFilipp Z, Zaid MA, Di Stasi A, Radojcic V, Betts CB, Coussens LM, Meyers ML, Qamoos H, Ordentlich P, Kumar V, Quaranto C, Schmitt A, Gu Y, Blazar BR, Wang TP, Salhotra A, Pusic I, Jagasia M, Lee SJ. Axatilimab for Chronic Graft-Versus-Host Disease After Failure of at Least Two Prior Systemic Therapies: Results of a Phase I/II Study. J Clin Oncol. 2023 Apr 1;41(10):1864-1875. doi: 10.1200/JCO.22.00958. Epub 2022 Dec 2. PMID 36459673

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Escalation: SNDX-6352 0.15 mg/kg Q2W: Participants received an intravenous (IV) infusion of SNDX-6352 0.15 milligrams (mg)/kilogram (kg) every 2 weeks (Q2W).
- Phase 1 Dose Escalation: SNDX-6352 0.5 mg/kg Q2W: Participants received an IV infusion of SNDX-6352 0.5 mg/kg Q2W.
- Phase 1 Dose Escalation: SNDX-6352 1 mg/kg Q2W; Phase 2 Dose Expansion: SNDX-6352 1 mg/kg Q2W: Participants received an IV infusion of SNDX-6352 1 mg/kg Q2W.
- Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q2W: Participants received an IV infusion of SNDX-6352 3 mg/kg Q2W.
- Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q4W: Participants received an IV infusion of SNDX-6352 3 mg/kg every 4 weeks (Q4W).
Period: Overall Study
Arm/Group | Phase 1 Dose Escalation: SNDX-6352 0.15 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 0.5 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 1 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q4W | Phase 2 Dose Expansion: SNDX-6352 1 mg/kg Q2W
Started | 1 | 1 | 3 | 6 | 7 | 23
Received at Least 1 Dose of Study Treatment | 1 | 1 | 3 | 6 | 6 | 23
Dose-limiting Toxicity (DLT) Evaluable (Participants who received at least one dose of SNDX-6352 were evaluated for DLTs over 2 cycles (Cycle 1 and Cycle 2).) | 1 | 1 | 3 | 6 | 6 | 0 (DLTs were not evaluated in Phase 2.)
Completed | 0 | 1 | 1 | 3 | 3 | 9
Not Completed | 1 | 0 | 2 | 3 | 4 | 14
Not completed — Investigator's Decision | 0 | 0 | 0 | 1 | 0 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Progressive Disease | 1 | 0 | 1 | 0 | 3 | 4
Not completed — Difficulty Coming into Site | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Drug Intolerance | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Noncompliance with follow-up visit | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Not Treated | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment.
Groups:
- Phase 1 Dose Escalation: SNDX-6352 0.15 mg/kg Q2W: Participants received an IV infusion of SNDX-6352 at 0.15 mg/kg Q2W.
- Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q4W: Participants received an IV infusion of SNDX-6352 3 mg/kg Q4W.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Escalation: SNDX-6352 0.15 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 0.5 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 1 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q4W | Phase 2 Dose Expansion: SNDX-6352 1 mg/kg Q2W | Total
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 6 | 23 | 40
Age, Continuous [Mean (Full Range); unit: years] | 64.0 [64 to 64] | 48.0 [48 to 48] | 43.7 [29 to 66] | 61.0 [53 to 73] | 59.2 [31 to 73] | 52.5 [16 to 69] | 54.7 [16 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 3 | 2 | 9 | 15
  Male | 1 | 1 | 2 | 3 | 4 | 14 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 3 | 6 | 6 | 22 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 1 | 0 | 0 | 1 | 1 | 2 | 5
  Race: White | 0 | 1 | 3 | 5 | 5 | 20 | 34
  Race: Other | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With DLTs
Description: A DLT was defined as the occurrence of any protocol-specified event within the first 28 days from the first dose of SNDX-6352 or administration of the third dose (Cycle 2 Day 1), whichever is later (from Cycle 1 Day 1 to Cycle 2 Day 1) and assessed by the Investigator as not being definitely attributable to underlying disease, disease progression, inter-current illness, concomitant medications or any other alternative cause.
Time Frame: Day 1 through the first 28 days from the first dose of SNDX-6352 or administration of the third dose (Cycle 2 Day 1), whichever is later (from Cycle 1 Day 1 to Cycle 2 Day 1)
Population: Participants who received at least 1 cycle of treatment and had at least one post-baseline response assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Dose Escalation: SNDX-6352 0.15 mg/kg: Participants received an IV infusion of SNDX-6352 0.15 mg/kg Q2W.
- Phase 1 Dose Escalation: SNDX-6352 0.5 mg/kg: Participants received an IV infusion of SNDX-6352 0.5 mg/kg Q2W.
- Phase 1 Dose Escalation: SNDX-6352 1 mg/kg: Participants received an IV infusion of SNDX-6352 1 mg/kg Q2W.
- Phase 1 Dose Escalation: SNDX-6352 3 mg/kg: Participants received an IV infusion of SNDX-6352 3 mg/kg Q2W.
Arm/Group | Phase 1 Dose Escalation: SNDX-6352 0.15 mg/kg | Phase 1 Dose Escalation: SNDX-6352 0.5 mg/kg | Phase 1 Dose Escalation: SNDX-6352 1 mg/kg | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 6
Participants | 0 | 0 | 0 | 2 | 0

2. Primary Outcome: Phase 1: Recommended Phase 2 Dose (RP2D)
Description: The RP2D was determined in discussion with the Sponsor, Medical Monitor, and Dose Determination Phase Investigators and was based on observations from the Phase 1 of the study (clinical benefit in chronic graft versus host disease [cGVHD] and pharmacokinetic/pharmacodynamic effects).
Time Frame: Day 1 through the first 28 days from the first dose of SNDX-6352 or administration of the third dose (Cycle 2 Day 1), whichever is later (from C1D1 to C2D1)
Population: Participants who received at least 1 cycle of treatment and had at least one post-baseline response assessment in Phase 1.
Measure: Number; unit: mg/kg
Groups:
- Phase 1 Dose Determination:SNDX-6352: Participants received an IV infusion of SNDX-6352 1 mg/kg Q2W.
Arm/Group | Phase 1 Dose Determination:SNDX-6352
Number analyzed (Participants) | 17
mg/kg | 1

3. Primary Outcome: Phase 2: Overall Response Rate (ORR) as Assessed by the Number of Participants With Complete Response (CR) or Partial Response (PR) at Cycle 7 Day 1 (Day 168)
Description: CR or PR was defined by the 2014 National Institutes of Health (NIH) Consensus Development Project on Criteria for Clinical Trials in cGVHD.CR was defined as resolution of all manifestations in each organ or site, and PR was defined as improvement in at least 1 organ or site without progression in any other organ or site. ORR was defined as the percentage of participants achieving a best overall response of CR or PR .ORR calculated as: (number of participants with best overall response as CR or PR)/total number of participants.
Time Frame: Cycle 7 Day 1 (Day 168)
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 Dose Expansion: SNDX-6352 1 mg/kg Q2W
Number analyzed (Participants) | 23
percentage of participants | 39.1 [19.71 to 61.46]

4. Secondary Outcome: Phase 1: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Measurable Concentration for SNDX-6352
Description: Blood samples were collected for determination of SNDX-6352 concentration.
Time Frame: Cycle 1: predose, at 30 min (end of infusion), and at 1 hour and 8 hours on Day 1 and Day 15
Population: Pharmacokinetic Analysis Set: All treated participants who had at least 1 plasma concentration measured. Number Analyzed = participants who were evaluable at specified timepoints
Measure: Mean (Full Range); unit: µg*h/mL
Groups:
- Phase 1 Dose Escalation: SNDX-6352 0.15 mg/kg Q2W: Participants received an IV infusion of SNDX-6352 0.15 mg/kg Q2W.
Arm/Group | Phase 1 Dose Escalation: SNDX-6352 0.15 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 0.5 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 1 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 6
µg*h/mL
  Cycle 1 Day 1 | 30.7 [30.7 to 30.7] | 96.2 [96.2 to 96.2] | 1546.0 [898.0 to 2140.0] | 10263.3 [4660.0 to 15300.0] | 12256.7 [6760.0 to 20700.0]
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 1 | 3 | 6 | 0
  Cycle 1 Day 15 | 22.9 [22.9 to 22.9] | 98.9 [98.9 to 98.9] | 714.0 [121.0 to 1740.0] | 14,055.0 [575.0 to 26,900.0] |

5. Secondary Outcome: Phase 1: Observed Maximum Plasma Concentration for SNDX-6352
Description: Blood samples were collected for determination of SNDX-6352 concentration.
Time Frame: Cycle 1: predose, at 30 min (end of infusion), and at 1 hour and 8 hours on Day 1 and Day 15
Population: as for outcome 4
Measure: Mean (Full Range); unit: µg/mL
Arm/Group | Phase 1 Dose Escalation: SNDX-6352 0.15 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 0.5 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 1 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 6
µg/mL
  Cycle 1 Day 1 | 4.6 [4.6 to 4.6] | 13.7 [13.7 to 13.7] | 26.7 [19.5 to 38.7] | 84.0 [63.0 to 106.0] | 82.2 [62.2 to 104.0]
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 1 | 3 | 6 | 0
  Cycle 1 Day 15 | 3.5 [3.5 to 3.5] | 14.2 [14.2 to 14.2] | 27.4 [20.1 to 41.3] | 91.8 [65.1 to 132.0] |

6. Secondary Outcome: Phase 1: Time to Observed Maximum Plasma Concentration
Description: Blood samples were collected for determination of SNDX-6352 concentration.
Time Frame: Cycle 1: predose, at 30 min (end of infusion), and at 1 hour and 8 hours on Day 1 and Day 15
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1 Dose Escalation: SNDX-6352 0.15 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 0.5 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 1 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 6
hours
  Cycle 1 Day 1 | 1.0 [1.0 to 1.0] | 1.5 [1.5 to 1.5] | 0.6 [0.6 to 0.6] | 0.9 [0.6 to 7.5] | 1.0 [0.5 to 7.9]
  Cycle 1 Day 15: number analyzed (Participants) | 1 | 1 | 3 | 6 | 0
  Cycle 1 Day 15 | 0.6 [0.6 to 0.6] | 0.5 [0.5 to 0.5] | 1.0 [0.6 to 1.5] | 1.0 [0.6 to 1.1] |

7. Secondary Outcome: Phase 1: Changes From Baseline in Colony-Stimulating Factor-1 (CSF-1) and Interleukin (IL-34) Serum Concentrations
Description: Blood samples were collected for determination of serum concentrations.
Time Frame: Baseline, Cycle 1 Day 8, Day 15, predose at Cycle 2 Day 1, Cycle 4 Day 1 (28-day cycles), and end of treatment (EOT) (median duration of treatment = 7 months)
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment. Number Analyzed = participants who were evaluable at specified timepoints
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Phase 1 Dose Escalation: SNDX-6352 0.15 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 0.5 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 1 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 6
pg/mL
  CSF-1 Cycle 1 Day 8 | 2.0 [2 to 2] | 602.0 [602 to 602] | 364480.0 [211185 to 400666] | 544837.5 [433627 to 613511] | 451482.0 [366543 to 697378]
  CSF-1 Cycle 1 Day 15: number analyzed (Participants) | 1 | 1 | 3 | 5 | 4
  CSF-1 Cycle 1 Day 15 | 69.0 [69 to 69] | -87.0 [-87 to -87] | 680.0 [-418 to 1556] | 897522.0 [75411 to 966627] | 821180.5 [581543 to 990015]
  CSF-1 Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 2 | 6
  CSF-1 Cycle 2 Day 1 | 19.0 [19 to 19] | 227.0 [227 to 227] | 400.0 [-126 to 60066] | 1474438.5 [1439355 to 1509522] | 773476.0 [11 to 1029015]
  CSF-1 Cycle 4 Day 1: number analyzed (Participants) | 0 | 1 | 3 | 2 | 2
  CSF-1 Cycle 4 Day 1 |  | 229.0 [229 to 229] | 465.0 [-319 to 1378480] | 899337.5 [-680 to 1799355] | 1386196.5 [603378 to 2169015]
  CSF-1 EOT: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  CSF-1 EOT | 63.0 [63 to 63] |  |  |  | 1709787.0 [1709787 to 1709787]
  IL-34 Cycle 1 Day 8 | 0 [0 to 0] | 0 [0 to 0] | 156.7 [86 to 409] | 576.2 [316 to 929] | 286.7 [81 to 775]
  IL-34 Cycle 1 Day 15: number analyzed (Participants) | 1 | 1 | 3 | 5 | 6
  IL-34 Cycle 1 Day 15 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 690.7 [199 to 1259] | 456.7 [216 to 744]
  IL-34 Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 2 | 6
  IL-34 Cycle 2 Day 1 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 42] | 1133.7 [979 to 1289] | 190.7 [0 to 931]
  IL-34 Cycle 4 Day 1: number analyzed (Participants) | 0 | 1 | 3 | 2 | 6
  IL-34 Cycle 4 Day 1 |  | 0 [0 to 0] | 0 [0 to 395] | 569.4 [0 to 1139] | 533.7 [241 to 827]
  IL-34 EOT: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
  IL-34 EOT | 0 [0 to 0] |  |  |  | 676.7 [676.7 to 676.7]

8. Secondary Outcome: Phase 1: Percent Change From Baseline in Nonclassical Monocytes (CD14+CD16++)
Description: Blood samples were collected for determination nonclassical monocytes levels.
Time Frame: Baseline, Day 8, Day 15, predose at Cycle 2 Day 1, Cycle 4 Day 1, and EOT (median duration of treatment = 7 months)
Population: as for outcome 7
Measure: Median (Full Range); unit: percent change
Arm/Group | Phase 1 Dose Escalation: SNDX-6352 0.15 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 0.5 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 1 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q4W
Number analyzed (Participants) | 0 | 1 | 2 | 5 | 6
percent change
  Cycle 1 Day 8 |  | -41.7 [-41.7 to -41.7] | -92.7 [-97 to -89] | -95.7 [-98 to -90] | -81.4 [-90 to -33]
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 1 | 2 | 4 | 4
  Cycle 1 Day 15 |  | -66.7 [-66.7 to -66.7] | 242.8 [-31 to 517] | -96.5 [-98 to -94] | -81.5 [-84 to 67]
  Cycle 1 Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 22 |  |  |  |  | -90.9 [-90.9 to -90.9]
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 1 | 1 | 1 | 6
  Cycle 2 Day 1 |  | -58.3 [-58.3 to -58.3] | -31.0 [-31.0 to -31.0] | -94.4 [-94.4 to -94.4] | -67.5 [-81 to 167]
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 1 | 2 | 2 | 2
  Cycle 4 Day 1 |  | -16.7 [-16.7 to -16.7] | 273.5 [41 to 506] | -76.5 [-99 to -54] | -82.5 [-91 to -74]
  EOT: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  EOT |  |  |  |  | -75.0 [-75.0 to -75.0]

9. Secondary Outcome: Phase 1: Number of Participants Positive for Anti-Drug Antibodies (ADA)
Description: Blood samples were collected for ADA assessment. A participant was considered ADA positive if at least 1 postbaseline sample was ADA positive.
Time Frame: Predose on Cycle 1 Day 1, Cycle 1 Day 15, Cycle 3 Day 1, Day 1 of each subsequent cycle through EOT plus 30 days after last dose (safety follow-up) (median duration of treatment = 7 months)
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Escalation: SNDX-6352 0.15 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 0.5 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 1 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q2W | Phase 1 Dose Escalation: SNDX-6352 3 mg/kg Q4W
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 6
Participants | 0 | 0 | 1 | 3 | 2

10. Secondary Outcome: Phase 2: Best Overall Response (BOR), as Defined by the 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD
Description: Physician-reported global cGVHD activity assessment and cGVHD response determination. Best overall response was calculated as percent of participants with a response of CR or PR.
Time Frame: Day 1 of each 28-Day cycle up to Cycle 7 Day 1
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 Dose Expansion: SNDX-6352 1 mg/kg Q2W
Number analyzed (Participants) | 23
percentage of participants | 78.3 [56.3 to 92.54]

11. Secondary Outcome: Phase 2: Failure Free Survival (FFS)
Description: FFS was defined as the time from first dose of study intervention to unequivocal progression of cGVHD or relapse of underlying malignancy or addition of another systemic immune suppressive therapy or discontinuation of study treatment due to toxicity or death for any reason. Unequivocal progression of cGVHD is defined as treatment discontinuation due to clinical progression. The duration of FFS was evaluated using organ-specific cGVHD activity assessment form and and summarized descriptively using the Kaplan-Meier method.
Time Frame: From first dose of study intervention (Day 1) up to 27 months
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Dose Expansion: SNDX-6352 1 mg/kg Q2W
Number analyzed (Participants) | 23
months | 16.9 [9.3 to NA] — The upper confidence interval (CI) was not evaluable due to insufficient number of participants with events.

12. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR was defined as the time of initial response until documented progression or start of another systemic treatment as assessed by the Kaplan-Meir method.
Time Frame: Day 1 of each 28-Day cycle for up to 12 cycles
Population: Participants who achieved PR or CR in the study were evaluable for DOR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2 Dose Expansion: SNDX-6352 1 mg/kg Q2W
Number analyzed (Participants) | 18
months | 9.53 [1.87 to 17.05]

13. Secondary Outcome: Phase 2: Sustained Response Rate (SRR)
Description: SSR of CR or PR ≥20 weeks was defined as rate of CR or PR lasting for at least 20 weeks from the time of initial response.
Time Frame: Day 1 of each 28-Day cycle for up to 12 cycles
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 Dose Expansion: SNDX-6352 1 mg/kg Q2W
Number analyzed (Participants) | 23
percentage of participants | 39.1 [19.7 to 61.5]

14. Secondary Outcome: Phase 2: Organ-specific Response Rate Based on 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD
Description: The percentage of participants with a response (CR/PR) in the skin, eyes, mouth, esophagus, upper gastrointestinal (GI), lower GI, liver, lungs, or joints and fascia were assessed using the NIH Consensus Development Project on Clinical Trials.
Time Frame: Day 1 of each 28-Day cycle for up to 12 cycles
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 Dose Expansion: SNDX-6352 1 mg/kg Q2W
Number analyzed (Participants) | 23
percentage of participants
  Esophagus: number analyzed (Participants) | 6
  Esophagus | 83.3 [35.88 to 99.58]
  Eyes: number analyzed (Participants) | 16
  Eyes | 18.8 [4.05 to 45.65]
  Joints and Fascia: number analyzed (Participants) | 17
  Joints and Fascia | 76.5 [50.1 to 93.19]
  Liver: number analyzed (Participants) | 3
  Liver | 0 [0 to 70.76]
  Lower GI: number analyzed (Participants) | 4
  Lower GI | 100.0 [39.76 to 100]
  Lungs: number analyzed (Participants) | 9
  Lungs | 33.3 [7.49 to 70.07]
  Mouth: number analyzed (Participants) | 12
  Mouth | 75.0 [42.81 to 94.51]
  Skin: number analyzed (Participants) | 21
  Skin | 19.0 [5.45 to 41.91]
  Upper GI: number analyzed (Participants) | 4
  Upper GI | 100.0 [39.76 to 100]
  Global | 47.8 [26.82 to 69.41]

15. Secondary Outcome: Phase 2: Number of Participants With a Joint and Fascia Response Based on Refined NIH Response Algorithm for cGVHD
Time Frame: Day 1 of each 28-Day cycle for up to 12 cycles
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment and who had this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Dose Expansion: SNDX-6352 1 mg/kg Q2W
Number analyzed (Participants) | 17
Participants
  Improved | 10
  Stable | 7

16. Secondary Outcome: Phase 2: Number of Participants With A Lee Symptom Scale Summary Score Decrease of at Least 7 Points From Baseline
Description: The Lee cGVHD symptom questionnaire asked participants to indicate the degree of "bother" that they experienced during the past 7 days due to symptoms in 7 domains potentially affected by chronic GVHD (skin, eyes and mouth, breathing, eating and digestion, muscles and joints, energy, emotional distress) using a 5-point Likert scale from 0 "not at all" to 4 "extremely." Scores were normalized (0 to 100 scale) and the number of participants with a ≥ 7-point decrease in normalized score was calculated. A decrease in score indicated improvement in symptoms.
Time Frame: Day 1 of each 28-Day cycle for up to 12 cycles
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Dose Expansion: SNDX-6352 1 mg/kg Q2W
Number analyzed (Participants) | 22
Participants | 12

17. Secondary Outcome: Phase 2: Number of Participants With a ≥50% Reduction in Prednisone Equivalent Dosage Lasting at Least 28 Days
Time Frame: Day 1 of each 28-Day cycle for up to 12 cycles
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment and had corticosteroid usage at Cycle 1 Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Dose Expansion: SNDX-6352 1 mg/kg Q2W
Number analyzed (Participants) | 19
Participants | 5

18. Secondary Outcome: Phase 2: Number of Participants Who Discontinued Calcineurin Inhibitor Use
Time Frame: Day 1 of each 28-Day cycle for up to 12 cycles
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment and had calcineurin inhibitors usage at Cycle 1 Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Dose Expansion: SNDX-6352 1 mg/kg Q2W
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to EOT plus 90 days after last dose (safety follow-up) (median duration of treatment = 7 months)
Description: Per pre-specified analysis, deaths and adverse events were collected by dose group. Therefore, data for participants who received dose group SNDX-6352 1 mg/kg Q2W in Phase 1 and Phase 2 are combined.
Groups:
- SNDX-6352 0.15 mg/kg Q2W: Participants received an IV infusion of SNDX-6352 0.15 mg/kg Q2W in Phase 1.
- SNDX-6352 0.5 mg/kg Q2W: Participants received an IV infusion of SNDX-6352 0.5 mg/kg Q2W in Phase 1.
- SNDX-6352 1 mg/kg Q2W: Participants received an IV infusion of SNDX-6352 1 mg/kg Q2W in Phases 1 and 2.
- SNDX-6352 3 mg/kg Q2W: Participants received an IV infusion of SNDX-6352 3 mg/kg Q2W in Phase 1.
- SNDX-6352 3 mg/kg Q4W: Participants received an IV infusion of SNDX-6352 3 mg/kg Q4W in Phase 1.
Arm/Group | SNDX-6352 0.15 mg/kg Q2W | SNDX-6352 0.5 mg/kg Q2W | SNDX-6352 1 mg/kg Q2W | SNDX-6352 3 mg/kg Q2W | SNDX-6352 3 mg/kg Q4W
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 1/26 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 12/26 | 3/6 | 2/6
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 26/26 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SNDX-6352 0.15 mg/kg Q2W (N=1) | SNDX-6352 0.5 mg/kg Q2W (N=1) | SNDX-6352 1 mg/kg Q2W (N=26) | SNDX-6352 3 mg/kg Q2W (N=6) | SNDX-6352 3 mg/kg Q4W (N=6)
Pneumonia (Infections and infestations) | 0 | 1 | 3 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Septic arthritis staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound infection pseudomonas (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Serratia sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SNDX-6352 0.15 mg/kg Q2W (N=1) | SNDX-6352 0.5 mg/kg Q2W (N=1) | SNDX-6352 1 mg/kg Q2W (N=26) | SNDX-6352 3 mg/kg Q2W (N=6) | SNDX-6352 3 mg/kg Q4W (N=6)
Fatigue (General disorders) | 0 | 1 | 12 | 3 | 2
Oedema peripheral (General disorders) | 1 | 0 | 4 | 1 | 2
Pyrexia (General disorders) | 0 | 0 | 2 | 3 | 0
Chills (General disorders) | 0 | 0 | 1 | 3 | 0
Malaise (General disorders) | 1 | 0 | 1 | 2 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 1 | 0
Oedema (General disorders) | 0 | 0 | 2 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 1 | 0
Axillary pain (General disorders) | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 6 | 4 | 4
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 3 | 6 | 5
Alanine aminotransferase increased (Investigations) | 1 | 0 | 5 | 4 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 4 | 4 | 3
Amylase increased (Investigations) | 1 | 0 | 6 | 4 | 0
Lipase increased (Investigations) | 0 | 0 | 4 | 3 | 3
Blood creatinine increased (Investigations) | 0 | 0 | 5 | 2 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 2 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 2 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 1 | 0
Blood creatine phosphokinase abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 1 | 0
C-reactive protein (Investigations) | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 0 | 1 | 0
Vitamin B1 decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 8 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 8 | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Tongue erythema (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 7 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Pustule (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound infection pseudomonas (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Abscess neck (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 3 | 2 | 3
Vision blurred (Eye disorders) | 0 | 0 | 3 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 2 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 2 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 2 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 6 | 3 | 1
Headache (Nervous system disorders) | 0 | 1 | 5 | 3 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 4 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 3 | 2 | 2
Haematoma (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urethral prolapse (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Androgen deficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT03604692/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT03604692/SAP_001.pdf